CLINICAL TRIAL: NCT01603550
Title: Brain Energy and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: United States Army Natick Soldier Research Development and Engineering Center (Unknown); Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Harris R. Lieberman, Research Psychologist, United States Army Research Institute of Environmental Medicine
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: H10-09
Record Dates: First submitted 2012-05-18; First posted 2012-05-23 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Energy Restriction; Sleep Deprivation
Keywords: energy restriction; sleep deprivation; cognitive performance; brain function
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Energy Restriction (Experimental)
  Interventions: Other: Energy Restriction
- Sleep Deprivation (Experimental)
  Interventions: Other: Sleep Deprivation

INTERVENTIONS:
Other: Sleep Deprivation — Sleep Deprivation
  Arms: Sleep Deprivation
Other: Energy Restriction — Energy Restriction
  Arms: Energy Restriction

SUMMARY:
This proposed laboratory study will extend previous findings on relationships between cognitive function and nutritional status to conditions that more closely resemble military operations where aerobic exercise, inadequate nutritional intake and sleep deprivation combine to degrade cognitive function. The investigators will examine cognitive function, brain activity and glucose levels in volunteers who are calorie-deprived, performing high workload cognitive tests, exercising and, in one arm of the study, are sleep-deprived for approximately 48 hours. A comprehensive cognitive test battery will be repeatedly administered and several cognitive tests will be administered when volunteers are exercising. Interstitial glucose levels will be assessed and whole body nitrogen utilization determined. The effects of energy restriction and the physiological basis of the relationship between peripheral glucose levels and cognitive function will be examined using a state-of-the-art imaging technology, functional Magnetic Resonance Imaging (fMRI). This technique will allow any key brain regions affected by caloric deprivation to be identified.

ELIGIBILITY:
Inclusion Criteria:

* MUST BE ACTIVE DUTY ARMY STATIONED AT NATICK SOLDIER SYSTEMS CENTER
* Fluent in English (non-native English speakers can be enrolled); males and females aged 18 - 39 years.

Exclusion Criteria:

* Not yet reached 18th birthday, metal implants - which can interfere with fMRI scanning; fear of small places; pregnant (USARIEM will test for pregnancy), Attention Deficit Hyperactivity Disorder (ADHD) - if previously documented by a waiver; acute or chronic physical limitation that would hinder performing cycle exercise; known allergies to medical adhesives.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harris R. Lieberman, PhD, Principal Investigator — US Army Research Institute of Environmental Medicine
Locations (1):
- USARIEM, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lieberman HR, Bukhari AS, Caldwell JA, Wilson MA, Mahoney CR, Pasiakos SM, McClung JP, Smith TJ. Two Days of Calorie Deprivation Induced by Underfeeding and Aerobic Exercise Degrades Mood and Lowers Interstitial Glucose but Does Not Impair Cognitive Function in Young Adults. J Nutr. 2017 Jan;147(1):110-116. doi: 10.3945/jn.116.238246. Epub 2016 Nov 2. PMID 27807037
- [Derived] Karl JP, Smith TJ, Wilson MA, Bukhari AS, Pasiakos SM, McClung HL, McClung JP, Lieberman HR. Altered metabolic homeostasis is associated with appetite regulation during and following 48-h of severe energy deprivation in adults. Metabolism. 2016 Apr;65(4):416-27. doi: 10.1016/j.metabol.2015.11.001. Epub 2015 Nov 6. PMID 26975533
- [Derived] O'Connor KL, Scisco JL, Smith TJ, Young AJ, Montain SJ, Price LL, Lieberman HR, Karl JP. Altered Appetite-Mediating Hormone Concentrations Precede Compensatory Overeating After Severe, Short-Term Energy Deprivation in Healthy Adults. J Nutr. 2016 Feb;146(2):209-17. doi: 10.3945/jn.115.217976. Epub 2016 Jan 6. PMID 26740683